CLINICAL TRIAL: NCT00115349
Title: Thalassemia Clinical Research Network - Cardiac L1/DFO Trial
Brief Title: Combination Therapy Compared With Single-Drug Therapy in Patients With Cardiac Diseases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to low enrollment
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 181; U01HL065260 (NIH); U01HL065244 (NIH); U01HL065239 (NIH); U01HL065238 (NIH); U01HL065232 (NIH)
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2014-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Beta-Thalassemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; beta-Thalassemia | interventions — Deferoxamine; Deferiprone; Long Interspersed Nucleotide Elements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L1/DFO (Experimental): Deferoxamine (DFO) and deferiprone (L1) combination therapy
  Interventions: Drug: Deferoxamine; Drug: Deferiprone (L1)
- DFO (Active Comparator): Deferoxamine (DFO) monotherapy
  Interventions: Drug: Deferoxamine

INTERVENTIONS:
Drug: Deferoxamine — Deferoxamine will be given daily for 12-24h/day 7 days a week either subcutaneous or intravenous at up to 50-60 mg/kg/day.
  Other Names: DFO
Drug: Deferiprone (L1) — The dose of L1, 75mg/kg in three divided oral doses, is the maximum dose at which toxicity has been tested in prospective trials
  Other Names: L1
  Arms: L1/DFO

SUMMARY:
The purpose of this study is to determine whether left ventricular function improves more rapidly with deferoxamine (DFO) and deferiprone (L1) combination therapy than with DFO monotherapy in patients with thalassemia and decreased ejection fractions. Secondary aims include evaluating changes in myocardial iron burden using T2* and estimating the relative incidence and severity of chelator-induced toxicity.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Participants will be randomized to 1 year of treatment with L1/DFO combination therapy or DFO monotherapy. At baseline, 6 months, and 1 year on therapy, cardiac function will be assessed by MRI measurement of left ventricular ejection fraction (LVEF), T2*, Holter monitoring, and electrocardiography. Additional monitoring for safety includes weekly blood testing, monthly visits, and periodic eye and ear exams.

ELIGIBILITY:
Inclusion Criteria:

* Transfusion-dependent beta-thalassemia (eight or more transfusion episodes in the previous year)
* Left ventricular ejection fraction by MRI less than or equal to 56% by balanced steady-state free precession (SSFP) or 63% by spoiled gradient recalled echo (SPGR)
* Currently on treatment with subcutaneous or intravenous DFO; participants must be willing and able to chelate 7 days per week 12 - 24 hours per day
* Serum ferritin greater than 1000 µg/L or ferritin between 500 µg/L and 1000 µg/L and cardiac T2* less than 20 ms

Exclusion Criteria:

* Pacemaker, severe claustrophobia, or other contraindications to MRI; severe congestive heart failure (New York Heart Association Classification IV); congenital or acquired valvular heart disease significant enough to require surgery or medications
* Currently receiving treatment for hepatitis; renal insufficiency defined by a clinically significant abnormal serum creatinine with a calculated creatinine clearance of less than 50 ml/min according to the Cockroft formula
* A neutrophil count less than 1.5 x 109/L on two or more occasions at least 4 weeks apart within the past year and not associated with an acute viral illness or a platelet count less than 80 x 109/L on two or more occasions at least 4 weeks apart within the past year
* Treatment with L1 or Exjade during the previous 2 weeks or previous adverse experience to L1 requiring suspension
* Infection with HIV
* Active participation in other investigational drug or device studies
* Unwilling to consider treatment with DFO at a dose of 50-60 mg/kg 12-24 hours per day 7 days per week
* Women who are pregnant or breast feeding
* Systemic infection or cardiovascular, hepatic, renal, pulmonary, or gastrointestinal disease that would prevent patients from undergoing any of the study-required treatments or procedures or requires treatment with any contraindicated medication(s)
* Presence of any other condition that, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with the patient's compliance with the protocol; may include but is not limited to alcohol or drug abuse
* For women of child-bearing potential, an inability or unwillingness to use a highly effective method of contraception (e.g., implants, injectables, combined oral contraceptives, or some intrauterine devices)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-06; Primary Completion 2008-07 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Porter, MD, Principal Investigator — University College, London; Patricia J. Giardina, MD, Study Chair — Weill Medical College of Cornell University; Ellis J. Neufeld, MD, Study Chair — Boston Children's Hospital; Elliott P, Vichinsky, MD, Study Chair — Children's Hospital and Research Institute, Oakland; Sonja McKinlay, Ph.D., Study Chair — New England Research Institutes, Inc.
Locations (6):
- United States (6):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital, Oakland, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital, Boston, Massachusetts
  - Weill Medical College of Cornell University, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled in August, 2005 and study closed due to low enrollment in June, 2008. 8 participating sites.
Pre-assignment Details: Patients were evaluated for eligibility based on the following criterial. If not eligible, they were not randomized to a treatment arm.
Groups:
- Deferoxamine (DFO) and Deferiprone (L1) Combination Therapy: DFO + L1 DFO Administered daily at 50-60 mg/kg for 12-24 hr/day 7 days a week either subcutaneous or intravenous.
  L1 Administered daily at 75 mg/kg in 3 divided doses taken orally and timed so that 2 of 3 doses will be simultaneous with DFO infusion.
- Deferoxamine (DFO) + Monotherapy: DFO + Placebo DFO Administered daily at 50-60 mg/kg for 12-24 hr/day 7 days a week either subcutaneous or intravenous.
  Placebo Administered orally three times daily.
Period: Overall Study
Arm/Group | Deferoxamine (DFO) and Deferiprone (L1) Combination Therapy | Deferoxamine (DFO) + Monotherapy
Started | 11 (Target was 43 subjects in this arm.) | 9 (Target was 43 subjects in this arm.)
Completed | 0 (Study closed due to low enrollment.) | 0 (study closed due to low enrollment.)
Not Completed | 11 | 9
Not completed — Study closed due to low enrollment. | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferoxamine (DFO) and Deferiprone (L1) Combination Therapy | Deferoxamine (DFO) + Monotherapy | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (5.1) | 25.8 (7.6) | 26.15 (6.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 3 | 6
  United States | 6 | 4 | 10
  Lebanon | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular Ejection Fraction (LVEF).
Description: The primary outcome variable is change in left ventricular ejection fraction (blood ejected from the heart into the body) as measured by MRI from baseline to one year. The unit of primary outcome (left ventricular ejection fraction) is the percent of the blood in left ventricle.
Time Frame: Baseline to one year
Measure: Least Squares Mean (Standard Error); unit: Percent of the blood in left ventricle
Arm/Group | Deferoxamine (DFO) and Deferiprone (L1) Combination Therapy | Deferoxamine (DFO) + Monotherapy
Number analyzed (Participants) | 11 | 9
Percent of the blood in left ventricle | 7.2 (1.9) | 6.3 (3.3)
Statistical Analysis 1: Comparison: Deferoxamine (DFO) and Deferiprone (L1) Combination Therapy vs Deferoxamine (DFO) + Monotherapy; The intended sample size of 86 patients (N=43 per arm) had 80% power to detect a 5% difference in LVEF between the two arms after 1 year of treatment, assuming a standard deviation of change in LVEF of 7.46%, and 20% loss to follow-up. The study was stopped early by NHLBI when analysis of the interim data confirmed a required sample size of 86 that was not achievable within the required time frame within the participating or planned centres; Test type: Superiority or Other; p = 0.89, Mixed Models Analysis; Linear mixed models with treatment, time, and treatment x time interaction were used, allowing for random participant-specific intercepts and slopes

2. Secondary Outcome: Evaluate Whether L1/DFO Combination Therapy is Superior to DFO Monotherapy in Lowering Myocardial Iron Burden Estimated by Myocardial T2*.
Time Frame: one year
Reporting Status: Not Posted

3. Secondary Outcome: Change in Left Ventricular (LV) Volume From Screening to One Year.
Time Frame: one year
Reporting Status: Not Posted

4. Secondary Outcome: Change in ECHO LV Volume, Ejection Fraction, Shortening Fraction, and VCFc/Wall Stress Z-score From Baseline to One Year.
Time Frame: one year
Reporting Status: Not Posted

5. Secondary Outcome: Change in Holter Monitor Scores From Baseline to One Year.
Time Frame: one year
Reporting Status: Not Posted

6. Secondary Outcome: Initiation of or Increase in Cardiac Medications
Time Frame: continuous
Reporting Status: Not Posted

7. Secondary Outcome: Adverse Events
Time Frame: continous
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Deferoxamine (DFO) and Deferiprone (L1) Combination Therapy | Deferoxamine (DFO) + Monotherapy
Serious Adverse Events (participants affected / at risk) | 6/11 | 3/9
Other Adverse Events (participants affected / at risk) | 8/11 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferoxamine (DFO) and Deferiprone (L1) Combination Therapy (N=11) | Deferoxamine (DFO) + Monotherapy (N=9)
Abnormal LFTs (Hepatobiliary disorders) | 1 (1) | 0 (0) — Nausea & abdominal discomfort occurring while taking deferiprone/placebo. Also reported "muscular type" aches & pains in the upper chest and arms. Severe elevation in liver enzymes was identified.
Congestive heart failure (Cardiac disorders) | 1 (1) | 2 (2) — Subject complaint of congestion and bloating. ECHO EF%= 20%, a decrease from 45%. Admitted for higher dose deferoxamine, & management. Deferoxamine was increased to 75 mg/kg/day, 7 days per week over 24 hours. Lasix 40 mg IV x 1 was administered.
Clot (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Pt had arm swelling and ultrasound revealed clot in left PICC line. Pt treated with vancomycin.
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) — Fever of 102 and cellulitis at the insertion site of his central venous catheter. Redness and pus drained from around this insertion site. The subject received nafcillin and Ceftriaxone IV. Desferal infusion continued during this time.
Meningitis (unkown viral vs. bacterial) (Infections and infestations) | 1 (1) | 0 (0) — Subject developed a fever 39.2C PO. Creatinine elevated to 2.2. Study drug held. CT without contrast done, "no obvious signs of meningitis or abcess." Treated w/ doses of Vancomycin and Cefotaxime.
Renal Disease (Renal and urinary disorders) | 1 (1) | 0 (0) — A routine chemistry showed elevated BUN 30mg/dl and creatinine 1.5mg/dl.
Palpitation (Cardiac disorders) | 0 (0) | 1 (2) — Subject complained of palpitations. ECG showed Atrial fibrillation. converting to normal sinus rhythm before started on any medication.
high grade fever and chills (Infections and infestations) | 1 (1) | 0 (0) — Subject complained of high grade fever and chills associated with dysuria. Subject presented to the ER and prelim results showed urinary tract infection but was admitted for monitoring due to low blood pressure.
Abdominal Pain (Hepatobiliary disorders) | 1 (1) | 0 (0) — Subject c/o stomach discomfort. 05/21 ANC was 1.4 and L1/Placebo was stopped. CBC was done and the ANC was 1.9. Treatment was restarted. An MRI (R2/T2*) was performed to assess liver iron. Summary stopped L1/Placebo, stopped DFO-S, MRI performed.
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Subject had been feeling fatigued with episodes of CP. Rx w/ Lasix and aldactone. Subject feeling worse with nausea and vomiting.CT scan showed left lower lobe pneumonia. Started on 10 day course of Levaquin. Discharged in good condition.
Splenectomy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Subject scheduled her for splenectomy. Had no complications.
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) — Subject admitted with CHF. Noted tachycardia to 140s. He was in atrial flutter, then atrial fibrillation. Was not hypotensive w/ no evidence of ventricular arrhythmia. Rx and converted to NSR. This event was possibly related to study drug.
Syncope (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Admitted with episode of syncope. His vision became dark and he felt dizzy. He was unable to support himself and fell to the ground hitting the side of his face. He reports that he was conscious throughout.
Watery diarrhea & hypotension (General disorders) | 1 (1) | 0 (0) — 5 day history of watery diarrhea. Dx w/ dehydration and syncopal event.
Retinal toxicity- drug induced (Eye disorders) | 1 (1) | 0 (0) — Distance vision was blurry and was seen by ophthalmology. ERG analysis shows deficits in both scotopic and photopic responses. These were not present on previous ERG. He c/o blurry vision and could not be corrected with glasses.
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Serum potassium =7.5 meq/L and received calcium carbonate infusion, and normal saline bolus. Glucose rose to 635 mg/dL. History of insulin dependent diabetes. Received Lasix & NS bolus were given. Potassium level returned to normal.
Central venous line infection (Infections and infestations) | 1 (2) | 0 (0) — Subject was admitted with cellulitis at the insertion site of his central venous catheter. The subject received vancomycin I.V. & developed Redman's syndrome. The vancomycin was stopped and was given Nafcillin IV.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferoxamine (DFO) and Deferiprone (L1) Combination Therapy (N=11) | Deferoxamine (DFO) + Monotherapy (N=9)
Abnormal LFTs (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bilerateral Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest Ache (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Common Cold (Social circumstances) | 1 (2) | 0 (0)
Dizziness (General disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epistaxis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fanconi (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 1 (1)
Kicked in chest (Social circumstances) | 1 (1) | 0 (0)
Low Grade Fever and Sore Throay (General disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Nausea and Vomiting (General disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (2)
Otitis media (Nervous system disorders) | 2 (2) | 0 (0)
Palpitations with dizziness (Cardiac disorders) | 1 (1) | 0 (0)
Phlebotic pain at blood infusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternocleidomastoid muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Strep Throat (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Vertigo (Vascular disorders) | 2 (2) | 0 (0)
Vomiting (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Allergic transfusion reactions hives (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
sore throat and cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
stomach flu (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
tooth ache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anxiety attack (Psychiatric disorders) | 0 (0) | 1 (2)
Heart palpatations (Cardiac disorders) | 0 (0) | 1 (1)
stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Shortness of Breath/fatigue (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ankle pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was stopped early by NHLBI when analysis of the interim data confirmed a required sample size of 86 that was not achievable within the required time frame within the participating or planned centres.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No